CLINICAL TRIAL: NCT00607854
Title: Safety and Efficacy of Ibritumomab Tiuxetan (Zevalin®) in Association With a Fludarabine Based Reduced Conditioning Regimen and Allogenic Stem Cell Support in Chemo-sensitive Relapsed CD20 Positive Aggressive Non-Hodgkin's Lymphoma Patients.
Brief Title: Safety of Ibritumomab Tiuxetan (Zevalin®) in Combination With a Fludarabine-based Reduced Intensity Conditioning (RIC) Regimen (ZEVALLO 2007)
Acronym: ZEVALLO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2007/11
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2013-02

CONDITIONS: Diffuse Large B-Cell Lymphoma; Mantle Cell Lymphoma
Keywords: Zevalin; Reduced intensity conditioning; Allogenic stem cell transplantation
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Mantle-Cell | interventions — ibritumomab tiuxetan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Zevalin (Experimental): Zevalin associated with a Fludarabine-based reduced-intensity conditioning regimen,all patients will receive Zevalin in the conditioning regimen
  Interventions: Drug: Ibritumomab Tiuxetan (Zevalin)

INTERVENTIONS:
Drug: Ibritumomab Tiuxetan (Zevalin) — Conditioning regimen followed by allogeneic hematopoietic stem cell transplantation.
  Ibritumomab Tiuxetan(Zevalin): 0.4 mCi/kg IV at day -14 (Day 0 is the transplantation)

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Zevalin® in a Reduced Intensity Conditioning regimen followed by allogenic stem cell support in patients with aggressive lymphomas who are responsive to a salvage chemotherapy regimen.

DETAILED DESCRIPTION:
The benefit of Zevalin® in the setting of autologous stem cell transplantation has been largely reported. The addition of Zevalin® to a fludarabine-based Reduced Intensity Conditioning regimen has been already evaluated in the setting of allo-SCT and the results reported so far seem to be promising without an overwhelming toxicity neither a delayed hematologic recovery. The assumption that the addition of Zevalin® to the conditioning regimen might improve lymphoma control and the demonstration that nucleoside analogs such as fludarabine synergize optimally with RIT led us to conduct this trial using the following preparative regimen: rituximab 250 mg/m² on days -21 and -14, Zevalin® 0,4 mCi/Kg body weight on day -14, fludarabine 30 mg/m² intravenously from days -6 to -2, Busulfan orally (4 mg/Kg body weight) or intravenously (0,8 mg/Kg body weight) on days -5 and -4 and ATG (Thymoglobulin®) 2,5 mg/Kg body weight intravenously on day -1. Cyclosporine A is administered at 2 or 3 mg/Kg body weight from day -1 to day 28 than followed by a dose reduction.

The purpose of this study is to evaluate the safety and efficacy of Zevalin® in a Reduced Intensity Conditioning regimen followed by allogenic stem cell support in patients with aggressive lymphomas who are responsive to a salvage chemotherapy regimen

Patients are followed from the beginning of the RIC regimen until day 365 for primary and secondary objectives of the study than on a regular basis depending on the practice of each centre. The evaluation includes physical examination (performance status, hematologic assessment, acute and chronic GVH disease), biologic tests (blood screening for blood count, renal and hepatic function, B and T-cell recovery, chimerism analysis, response assessment) and complementary examinations (marrow biopsies, tomography scan, positron emission tomography, …).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 65
* Patients with this lymphoma:

  1. CD20 positive diffuse large B-cell lymphoma in relapse or refractory after two prior regimens or after one regimen including autologous stem cell transplantation, or
  2. CD20 positive mantle-cell lymphoma in relapse or refractory after two prior regimens or after one regimen including autologous stem cell transplantation or
  3. Other CD20 positive aggressive lymphoma for which an indication of allograft is selected (Burkitt lymphoma, lymphoblastic lymphoma, intra-vascular lymphoma…..) or
  4. Low grade lymphoma CD20 positive (follicular lymphoma, marginal zone lymphoma) in histological processing or
  5. Low grade lymphoma CD20 positive for which an indication of allograft is selected
* And sensitive to relapse's treatment
* HLA-matched related or unrelated donor 10/10 or 9/10 with C or DQ mismatch without contra-indication for stem cell mobilization
* ECOG (Eastern Cooperative Oncology Group) < 2
* Having or not received previously rituximab
* With a chemosensitive relapse NHL (at least partial response > 50% as defined with cheson criteria (See appendix 5)
* Eligible for an allogenic transplant
* With a signed informed consent (obtained on the screening day at the latest and before any investigation)
* Patient affiliated to or beneficiary of the National Health Service

Exclusion Criteria:

* Patient allografted previously
* History of cancer
* Patient with HIV or HCV positive serology and requiring treatment
* Childbearing or child breastfeeding women
* Women who are pregnant or nursing, or man, in the absence of effective contraception during treatment and up to 12 months after stopping treatment
* Any contraindication to allogenic stem cell transplantation:
* Cardiac insufficiency (ejection fraction < 50% by echocardiography)
* Respiratory insufficiency defined as DLCO below 50% of the theoretical value
* Renal failure defined as creatinin clearance < 30 ml/mn
* Hepatic failure defined as a 2-fold increase of bilirubin or transaminases except if due to the lymphoma
* Known hypersensitivity to murine antibodies and other proteins, the active ingredients or any of the ingredients of the products under review
* Patient under the protection of justice

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-02; Primary Completion 2011-02 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
the treatment-related mortality rate (except if the death is related to the lymphoma exclusively). | day 100 post transplant

SECONDARY OUTCOMES:
The event-free-survival (EFS)(an event is defined as: death from any cause, relapse or progression, need to another treatment except for donor-lymphocytes injection (DLI), patient lost for follow-up) | 1 year post transplant
The rate of hematologic recovery (defined as ANC above 500/mm3 and platelets count above 20.000/mm3 for three consecutive days without stimulating growth support neither platelet transfusion) | day 30
Biological post allogenic effects of Zevalin® on the incidence of GVHD and B-cell and T-cell reconstitution | days d0, d28, d90, d180 and 1 year
Chimérism | day d28, d56, d 80, 1 year than at least once a year

CONTACTS AND LOCATIONS:
Overall Officials: Krimo BOUABDALLAH, MD, Principal Investigator — University Hospital Bordeaux, France; Geneviève CHENE, Pr, Study Chair — University Hospital Bordeaux, France
Locations (12):
- France (12):
  - Service d'hématologie - CHU de Besançon, Besançon
  - Service des maladies du sang - Hôpital Haut-Lévêque - avenue de magellan, Bordeaux - Pessac
  - Service d'hématologie - CHU Hôtel Dieu Clermont-Ferrand, Clermont-Ferrand
  - Service de médecine nucléaire - Centre de Lutte contre le Cancer de la Région Auvergne Jean Perrin, Clermont-Ferrand
  - Hôpital Edouard Herriot, Lyon
  - Service d'Oncologie Hématologie, Institut Paoli Calmettes - 232 Bd Ste Marguerite, Marseille
  - Hématologie et Oncologie médicale - CHU Lapeyronie, Montpellier
  - Service d'Hématologie, Hôpital Hôtel Dieu, CHU Nantes - 1 Place Alexis Ricordeau, Nantes
  - Service d'hématologie clinique - Hôpital l'Archet 1, Nice
  - Service d'Hématologie Adultes - Hôpital Necker-Enfants Malade, Paris
  - Pôle hématologie et immunologie clinique - Hôpital Saint-Louis, Paris
  - Département d'hématologie et d'Oncologie - CHRU Hautepierre, Strasbourg

REFERENCES:
- [Background] Cheson BD. The role of radioimmunotherapy with yttrium-90 ibritumomab tiuxetan in the treatment of non-Hodgkin lymphoma. BioDrugs. 2005;19(5):309-22. doi: 10.2165/00063030-200519050-00004. PMID 16207072
- [Background] Chopra R, Goldstone AH, Pearce R, Philip T, Petersen F, Appelbaum F, De Vol E, Ernst P. Autologous versus allogeneic bone marrow transplantation for non-Hodgkin's lymphoma: a case-controlled analysis of the European Bone Marrow Transplant Group Registry data. J Clin Oncol. 1992 Nov;10(11):1690-5. doi: 10.1200/JCO.1992.10.11.1690. PMID 1403052
- [Background] Dean RM, Fowler DH, Wilson WH, Odom J, Steinberg SM, Chow C, Kasten-Sportes C, Gress RE, Bishop MR. Efficacy of reduced-intensity allogeneic stem cell transplantation in chemotherapy-refractory non-hodgkin lymphoma. Biol Blood Marrow Transplant. 2005 Aug;11(8):593-9. doi: 10.1016/j.bbmt.2005.04.005. PMID 16041309
- [Background] Escalon MP, Champlin RE, Saliba RM, Acholonu SA, Hosing C, Fayad L, Giralt S, Ueno NT, Maadani F, Pro B, Donato M, McLaughlin P, Khouri IF. Nonmyeloablative allogeneic hematopoietic transplantation: a promising salvage therapy for patients with non-Hodgkin's lymphoma whose disease has failed a prior autologous transplantation. J Clin Oncol. 2004 Jun 15;22(12):2419-23. doi: 10.1200/JCO.2004.09.092. PMID 15197204
- [Background] Fietz T, Uharek L, Gentilini C, Muessig A, Rieger K, Marinets O, Sandrock D, Munz DL, Glass B, Thiel E, Blau IW. Allogeneic hematopoietic cell transplantation following conditioning with 90Y-ibritumomab-tiuxetan. Leuk Lymphoma. 2006 Jan;47(1):59-63. doi: 10.1080/10428190500260478. PMID 16321828
- [Background] Frater JL, Hsi ED. Properties of the mantle cell and mantle cell lymphoma. Curr Opin Hematol. 2002 Jan;9(1):56-62. doi: 10.1097/00062752-200201000-00010. PMID 11753079
- [Background] Freytes CO, Loberiza FR, Rizzo JD, Bashey A, Bredeson CN, Cairo MS, Gale RP, Horowitz MM, Klumpp TR, Martino R, McCarthy PL, Molina A, Pavlovsky S, Pecora AL, Serna DS, Tsai T, Zhang MJ, Vose JM, Lazarus HM, van Besien K; Lymphoma Working Committee of the International Bone Marrow Transplant Registry. Myeloablative allogeneic hematopoietic stem cell transplantation in patients who experience relapse after autologous stem cell transplantation for lymphoma: a report of the International Bone Marrow Transplant Registry. Blood. 2004 Dec 1;104(12):3797-803. doi: 10.1182/blood-2004-01-0231. Epub 2004 Jul 27. PMID 15280203
- [Background] Gianni AM, Cortelazzo S, Magni M, Martelli M; Michelangelo Cooperative. Rituximab: enhancing stem cell transplantation in mantle cell lymphoma. Bone Marrow Transplant. 2002 Feb;29 Suppl 1:S10-3. doi: 10.1038/sj.bmt.1703296. PMID 11840155
- [Background] Gopal AK, Pagel JM, Rajendran JG, Maloney DG, Appelbaum FR, Sorror ML, Sandmaier BM, Storb R, Press OW. Improving the efficacy of reduced intensity allogeneic transplantation for lymphoma using radioimmunotherapy. Biol Blood Marrow Transplant. 2006 Jul;12(7):697-702. doi: 10.1016/j.bbmt.2006.03.014. PMID 16785058
- [Background] Grigg A, Ritchie D. Graft-versus-lymphoma effects: clinical review, policy proposals, and immunobiology. Biol Blood Marrow Transplant. 2004 Sep;10(9):579-90. doi: 10.1016/j.bbmt.2004.05.008. PMID 15319770
- [Background] Haioun C, Lepage E, Gisselbrecht C, Salles G, Coiffier B, Brice P, Bosly A, Morel P, Nouvel C, Tilly H, Lederlin P, Sebban C, Briere J, Gaulard P, Reyes F. Survival benefit of high-dose therapy in poor-risk aggressive non-Hodgkin's lymphoma: final analysis of the prospective LNH87-2 protocol--a groupe d'Etude des lymphomes de l'Adulte study. J Clin Oncol. 2000 Aug;18(16):3025-30. doi: 10.1200/JCO.2000.18.16.3025. PMID 10944137
- [Background] Johnson TA, Press OW. Synergistic cytotoxicity of iodine-131-anti-CD20 monoclonal antibodies and chemotherapy for treatment of B-cell lymphomas. Int J Cancer. 2000 Jan 1;85(1):104-12. doi: 10.1002/(sici)1097-0215(20000101)85:13.0.co;2-g. PMID 10585592
- [Background] Jones RJ, Ambinder RF, Piantadosi S, Santos GW. Evidence of a graft-versus-lymphoma effect associated with allogeneic bone marrow transplantation. Blood. 1991 Feb 1;77(3):649-53. PMID 1991174
- [Background] Khouri IF, Keating M, Korbling M, Przepiorka D, Anderlini P, O'Brien S, Giralt S, Ippoliti C, von Wolff B, Gajewski J, Donato M, Claxton D, Ueno N, Andersson B, Gee A, Champlin R. Transplant-lite: induction of graft-versus-malignancy using fludarabine-based nonablative chemotherapy and allogeneic blood progenitor-cell transplantation as treatment for lymphoid malignancies. J Clin Oncol. 1998 Aug;16(8):2817-24. doi: 10.1200/JCO.1998.16.8.2817. PMID 9704734
- [Background] Khouri IF, Lee MS, Romaguera J, Mirza N, Kantarjian H, Korbling M, Albitar M, Giralt S, Samuels B, Anderlini P, Rodriguez J, von Wolff B, Gajewski J, Cabanillas F, Champlin R. Allogeneic hematopoietic transplantation for mantle-cell lymphoma: molecular remissions and evidence of graft-versus-malignancy. Ann Oncol. 1999 Nov;10(11):1293-9. doi: 10.1023/a:1008380527502. PMID 10631455
- [Background] Khouri IF, Lee MS, Saliba RM, Jun G, Fayad L, Younes A, Pro B, Acholonu S, McLaughlin P, Katz RL, Champlin RE. Nonablative allogeneic stem-cell transplantation for advanced/recurrent mantle-cell lymphoma. J Clin Oncol. 2003 Dec 1;21(23):4407-12. doi: 10.1200/JCO.2003.05.501. PMID 14645431
- [Background] Maris MB, Sandmaier BM, Storer BE, Chauncey T, Stuart MJ, Maziarz RT, Agura E, Langston AA, Pulsipher M, Storb R, Maloney DG. Allogeneic hematopoietic cell transplantation after fludarabine and 2 Gy total body irradiation for relapsed and refractory mantle cell lymphoma. Blood. 2004 Dec 1;104(12):3535-42. doi: 10.1182/blood-2004-06-2275. Epub 2004 Aug 10. PMID 15304387
- [Background] Milpied N, Deconinck E, Gaillard F, Delwail V, Foussard C, Berthou C, Gressin R, Lucas V, Colombat P, Harousseau JL; Groupe Ouest-Est des Leucemies et des Autres Maladies du Sang. Initial treatment of aggressive lymphoma with high-dose chemotherapy and autologous stem-cell support. N Engl J Med. 2004 Mar 25;350(13):1287-95. doi: 10.1056/NEJMoa031770. PMID 15044639
- [Background] Morris E, Thomson K, Craddock C, Mahendra P, Milligan D, Cook G, Smith GM, Parker A, Schey S, Chopra R, Hatton C, Tighe J, Hunter A, Peggs K, Linch D, Goldstone A, Mackinnon S. Outcomes after alemtuzumab-containing reduced-intensity allogeneic transplantation regimen for relapsed and refractory non-Hodgkin lymphoma. Blood. 2004 Dec 15;104(13):3865-71. doi: 10.1182/blood-2004-03-1105. Epub 2004 Aug 10. PMID 15304395
- [Background] Nademanee A, Forman SJ. Role of hematopoietic stem cell transplantation for advanced-stage diffuse large cell B-cell lymphoma-B. Semin Hematol. 2006 Oct;43(4):240-50. doi: 10.1053/j.seminhematol.2006.07.006. PMID 17027658
- [Background] Philip T, Guglielmi C, Hagenbeek A, Somers R, Van der Lelie H, Bron D, Sonneveld P, Gisselbrecht C, Cahn JY, Harousseau JL, et al. Autologous bone marrow transplantation as compared with salvage chemotherapy in relapses of chemotherapy-sensitive non-Hodgkin's lymphoma. N Engl J Med. 1995 Dec 7;333(23):1540-5. doi: 10.1056/NEJM199512073332305. PMID 7477169
- [Background] Ratanatharathorn V, Uberti J, Karanes C, Abella E, Lum LG, Momin F, Cummings G, Sensenbrenner LL. Prospective comparative trial of autologous versus allogeneic bone marrow transplantation in patients with non-Hodgkin's lymphoma. Blood. 1994 Aug 15;84(4):1050-5. PMID 8049425
- [Background] Reyes F, Lepage E, Ganem G, Molina TJ, Brice P, Coiffier B, Morel P, Ferme C, Bosly A, Lederlin P, Laurent G, Tilly H; Groupe d'Etude des Lymphomes de l'Adulte (GELA). ACVBP versus CHOP plus radiotherapy for localized aggressive lymphoma. N Engl J Med. 2005 Mar 24;352(12):1197-205. doi: 10.1056/NEJMoa042040. PMID 15788496
- [Background] Rodriguez R, Nademanee A, Ruel N, Smith E, Krishnan A, Popplewell L, Zain J, Patane K, Kogut N, Nakamura R, Sarkodee-Adoo C, Forman SJ. Comparison of reduced-intensity and conventional myeloablative regimens for allogeneic transplantation in non-Hodgkin's lymphoma. Biol Blood Marrow Transplant. 2006 Dec;12(12):1326-34. doi: 10.1016/j.bbmt.2006.08.035. PMID 17162215
- [Background] Schimmer AD, Jamal S, Messner H, Keating A, Meharchand J, Huebsch L, Walker I, Benger A, Gluck S, Smith A. Allogeneic or autologous bone marrow transplantation (BMT) for non-Hodgkin's lymphoma (NHL): results of a provincial strategy. Ontario BMT Network, Canada. Bone Marrow Transplant. 2000 Oct;26(8):859-64. doi: 10.1038/sj.bmt.1702625. PMID 11081385
- [Background] Shenkier TN, Voss N, Fairey R, Gascoyne RD, Hoskins P, Klasa R, Klimo P, O'Reilly SE, Sutcliffe S, Connors JM. Brief chemotherapy and involved-region irradiation for limited-stage diffuse large-cell lymphoma: an 18-year experience from the British Columbia Cancer Agency. J Clin Oncol. 2002 Jan 1;20(1):197-204. doi: 10.1200/JCO.2002.20.1.197. PMID 11773170
- [Background] Slavin S, Nagler A, Naparstek E, Kapelushnik Y, Aker M, Cividalli G, Varadi G, Kirschbaum M, Ackerstein A, Samuel S, Amar A, Brautbar C, Ben-Tal O, Eldor A, Or R. Nonmyeloablative stem cell transplantation and cell therapy as an alternative to conventional bone marrow transplantation with lethal cytoreduction for the treatment of malignant and nonmalignant hematologic diseases. Blood. 1998 Feb 1;91(3):756-63. PMID 9446633
- [Background] Vandenberghe E, Ruiz de Elvira C, Loberiza FR, Conde E, Lopez-Guillermo A, Gisselbrecht C, Guilhot F, Vose JM, van Biesen K, Rizzo JD, Weisenburger DD, Isaacson P, Horowitz MM, Goldstone AH, Lazarus HM, Schmitz N. Outcome of autologous transplantation for mantle cell lymphoma: a study by the European Blood and Bone Marrow Transplant and Autologous Blood and Marrow Transplant Registries. Br J Haematol. 2003 Mar;120(5):793-800. doi: 10.1046/j.1365-2141.2003.04140.x. PMID 12614212
- [Background] Winter JN. Combining yttrium 90-labeled ibritumomab tiuxetan with high-dose chemotherapy and stem cell support in patients with relapsed non-Hodgkin's lymphoma. Clin Lymphoma. 2004 Oct;5 Suppl 1:S22-6. doi: 10.3816/clm.2004.s.005. PMID 15498146
- [Derived] Bouabdallah K, Furst S, Asselineau J, Chevalier P, Tournilhac O, Ceballos P, Vigouroux S, Tabrizi R, Doussau A, Bouabdallah R, Mohty M, Le Gouill S, Blaise D, Milpied N. 90Y-ibritumomab tiuxetan, fludarabine, busulfan and antithymocyte globulin reduced-intensity allogeneic transplant conditioning for patients with advanced and high-risk B-cell lymphomas. Ann Oncol. 2015 Jan;26(1):193-198. doi: 10.1093/annonc/mdu503. Epub 2014 Oct 30. PMID 25361987